CLINICAL TRIAL: NCT01158495
Title: Differentiating Outcome Measures in Infant and Early Childhood Lung Disease Utilizing Controlled Ventilation Infant/Young Child Chest CT Scanning and Lung Function Testing
Brief Title: Outcome Measures in Infant/Early Childhood Lung Disease w/ Chest CT Scanning & Lung Function Testing
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSVAR0009; SU-07062010-6488 (Other: Stanford University)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Intubation with a cuffed ET Tube
Procedure: CT scan Radiation

SUMMARY:
To implement a new method of performing chest CT imaging in young children at Packard Children's Hospital entitled controlled ventilation infant/young child chest CT scanning. This technique will be used to evaluate early lung disease comparing quantitative chest CT air trapping and airway measurements with lung function measurements in infants, toddlers, and young children with chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:1) Infants and young children (age <= 3 months to < 5 years) and either 2) or 3) below.

2) Respiratory condition (e.g. cystic fibrosis (CF), primary ciliary dyskinesia, bronchopulmonary dysplasia, asthma, or other pulmonary condition) and under the care of a pediatric pulmonologist at LPCH.

3) Oncology condition (e.g. young children with or without cancer, who are being screened for lung metastasis) and are being followed by pediatric oncologists at LPCH.

4) For minors, informed consent by parent or legal guardian.

5) Ability to comply with study visit procedures as judged by the investigator. Exclusion Criteria:1) Acute wheezing and/or respiratory distress at Study visit.

2) Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset in 1 week preceding Study visit.

3) Oxygen saturation < 90% on room air at study visit.

4) Any medical condition that in the opinion of the investigator precludes subject participation.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants/young children with cystic fibrosis, primary ciliary dyskinesia, or other chronic lung disease, followed at our CF Center or Pulmonary Clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Quantitative CT air trapping & airway measurements | 6 mo

SECONDARY OUTCOMES:
Functional residual capacity (FRC) & Lung Clearance Index (LCI). | 6 mo
Differences between Quantitative CT air trapping & airway measurements & multibreath washout (MBW) FRC and LCI. | 6 mo
Correlation between LCI and quantitative air trapping | 6 mo
Correlation between bronchial wall thickness measurements/bronchiectasis measurements and LCI/FRC | 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Terry Earl Robinson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States